CLINICAL TRIAL: NCT05212961
Title: Clinical Profile and Outcome of Post Covid-19 Rhino-orbital Fungal Mucormycosis in Minia Governorate
Brief Title: COVID-19 and Rhino-orbital Mucormycosis
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sahar T A Abdelaziz, Assistant Professor, Minia University
Other Study IDs: Ophthalmology
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Mucormycosis
MeSH Terms: conditions — Mucormycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detect the clinical presentation and outcome of post covid-19 fungal mucormycosis in patients referred to Minia university Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had positive PCR test for Covid-19.
2. Fungal rhino-orbital infection was confirmed.

Exclusion Criteria:

1. Suspected patient with COVID-19 not confirmed with PCR
2. Incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had fungal rhino-orbital infection and positive PCR test for Covid-19. was confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Outcome of rhino-orbital mucormycosis in COVID-19 patients | 9 months
  Data of the patients who had post Covid-19 fungal mucormycosis in the last year will be revised to detect clinical presentation and final outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Minia University, Minya, Egypt